CLINICAL TRIAL: NCT04405310
Title: Plasma From Covalescent Donors With Covid-19 for the Management of Patients With SARS-COV-2 Fase II and III, a Doble Center Randomized Doble Blind Trial
Brief Title: Convalescent Plasma of Covid-19 to Treat SARS-COV-2 a Randomized Doble Blind 2 Center Trial
Acronym: CPC-SARS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Mexicano para el Estudio de la Medicina Intensiva (Other)
Collaborators: Hospital General Naval de Alta Especialidad - Escuela Medico Naval (Other Government); National Institute of Pediatrics, Mexico (Other Government); Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Angel Augusto Perez Calatayud, Head of division of critical care, Grupo Mexicano para el Estudio de la Medicina Intensiva
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DI/20/201/04/19
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: SARS Pneumonia
Keywords: SARS-COV-2, CONVALESCENT PLASMA

STUDY DESIGN:
Intervention Model Description: Parallel assignment, relationship 3.2.3
Who Masked: Participant, Care Provider
Masking Description: parallel design 3:2:3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- EXP-PC-F2 (Experimental): Patients with Pneumonia due to SARS-COV-2 phase 2 with Hyperimmune Plasma from Convalescent patients and conventional Therapy (Azithromycin and Hydroxychloroquine)
  Interventions: Biological: Convalescent Plasma of patients with COVID-19
- EXP-NONPC-F2 (Placebo Comparator): 20 Patients with Pneumonia due to SARS-COV-2 phase 2 with conventional Therapy (Azithromycin and Hydroxychloroquine) and 20% Albumin in Hartman Solution.
  Interventions: Other: placebo (hartmann plus albumine)
- EXP-PC-F3 (Experimental): 20 Patients with Pneumonia due to SARS-VOC-2 phase 3 with Hyperimmune Plasma from Convalescent patients and conventional Therapy (Azithromycin and Hydroxychloroquine)
  Interventions: Biological: Convalescent Plasma of patients with COVID-19
- EXP-NONPC-F3 (Placebo Comparator): 20 Patients with Pneumonia due to SARS-VOC-2 phase 3 with conventional Therapy (Azithromycin and Hydroxychloroquine) and 20% Albumin in Hartman Solution.
  Interventions: Other: placebo (hartmann plus albumine)

INTERVENTIONS:
Biological: Convalescent Plasma of patients with COVID-19 — Convalescent Plasma from patients with covid-19 by Apheresis, the maximum plasma volume withdrawn per session should not exceed 600 mL, excluding the anticoagulant volume, or 16% of the total blood volume, in the absence of volumetric replacement.
  Other Names: Hyperinmunne plasma
  Arms: EXP-PC-F2; EXP-PC-F3
Other: placebo (hartmann plus albumine) — use of albumin 20% in 250cc of Hartmann solution
  Arms: EXP-NONPC-F2; EXP-NONPC-F3

SUMMARY:
The new SARS-CoV-2 coronavirus is an emerging virus originating in Wuhan, China that has spread rapidly throughout the world. As of March 24, 2020, China had reported 81,767 cases with 3,281 deaths, and the World Health Organization (WHO) declared coronavirus 19 (COVID-19) a pandemic. COVID-19 disease is currently a pandemic without specific therapeutic agents and substantial mortality. So it is of utmost importance to find new treatments. Various therapies, such as Remdesivir and Favipiravir, are being investigated but the antiviral efficacy of these drugs is not yet known. The use of convalescent plasma was used as an empirical treatment during the Ebola virus outbreaks in 2014 and in 2015 a protocol was established for the treatment of the Middle East respiratory syndrome coronavirus (MERS) with convalescent plasma. This approach with other viral infections such as SARS-CoV, H5N1 avian influenza and H1N1 influenza suggesting that plasma transfusion from convalescent donors was effective.

For this study, plasma from convalescent donors will be collected from those donors who have recovered from SARS-CoV-2 and are between 10 and 14 days after illness. Immunoassays will be carried out to detect total IgM and IgG antibodies against SARS-CoV-2. Patients will receive 1 to 3 convalescent plasma transfusions, depending on the response to treatment.

The expected results are: normal body temperature, decrease in viral load or negative between 10-12 days after transfusion of convalescent plasma, which does not progress to ARDS, extubation of mechanical ventilation within two weeks of treatment, recovery of patient.

DETAILED DESCRIPTION:
Currently, SARS-CoV-2 disease represents a Public Health emergency of international concern. The new coronavirus COVID-19 is estimated to have infected more than 1.8 million people worldwide. The WHO estimates that the contagion rate (R0) of the virus is 1.4 to 2.5, which affects its exponential replication. In the absence of an effective treatment for SARS-CoV-2 disease, there is an urgent need to evaluate therapeutic alternatives that reduce the mortality and morbidity of this virus. There is scientific evidence that supports the use of convalescent donor plasma for the treatment of emerging virus outbreaks and suggests that the transfusion of convalescent donor plasma is effective, and therefore the following question is established:

The use of plasma from convalescent donors by COVID-19 in patients with SARS-CoV-2 disease, stage II (moderate) and III (severe), is a treatment that reduces mortality?

Given that the mortality rate is a very relevant fact, which concerns the general population, the clinical treatments that can be used to reduce the mortality rate of critical cases are of great relevance. There are patients recovered from COVID-19 who are potential plasma donors, and in turn, many critical patients who need to receive it.

Currently, there are no effective treatments to address COVID-19 disease. A recent WHO report indicates that early results with the use of convalescent plasma suggest that it may be a potentially useful treatment modality for severe SARS-CoV-2 disease. The use of convalescent plasma from COVID-19 in acute infected patients is currently considered an experimental therapy. This implies the need to promote clinical trials in order to demonstrate their efficacy. It is recommended that the entire process from donor selection, processing, labeling, storage and distribution to be carried out in a specifically licensed institution. These institutions must have all the guarantees that prove the correct practice of the procedures.

The use of convalescent plasma has been used as rescue therapy in patients with SARS whose condition continues to deteriorate despite treatment with methylprednisolone pulses, in addition, different studies have shown a decrease in hospital stay, and lower mortality in patients treated with convalescent plasma compared to those in which this treatment was not used.

A multicenter randomized study by Hung showed that the use of convalescent plasma in patients with type A H1N1 influenza was associated with a lower viral load and a reduction in mortality 5 days after the onset of symptoms. A Mair-Jenkins meta-analysis showed that mortality was reduced after several doses of convalescent plasma, and another meta-analysis by Luke identified in 1703 patients with influenza pneumonia (1918-1925) that the use of convalescent plasma blood products an absolute reduction. 21% (95% CI 15-27; p = 0.001) in crude fatality with low risk of bias.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 70 years of age.
* Serious or critically ill patients confirmed for SARS-CoV-2 disease (RT-PCR).
* Meet the criteria for Disease with SARS-CoV-2 disease, phase II (Moderate) and phase III (severe) .
* Suspected Cytokine Release Syndrome with Hscore 169 points.
* Presence of severe acute hypoxemia with SpO2 <90% in ambient air and / or PaO2 / FiO2 <300 mmHg.
* Meet criteria (plain chest tomography or plain chest radiograph) for SARS-CoV-2 disease.
* Supplemental oxygen requirement either through the facial store plus reservoir bag, high-flow nasal tips or advanced airway management and invasive mechanical ventilation support.

Exclusion Criteria:

* patient has no interest in participating in the trial.
* Bilateral pulmonary infiltrate related to heart failure or other cause of water overload.
* Virus positive respiratory viral panel other than COVID-19
* History of allergy to plasma, sodium citrate, or methylene blue.
* Patients with a history of autoimmune diseases or selective IgA insufficiency.
* Those patients who are participating in other protocols.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Death | 15 days
  any cause

SECONDARY OUTCOMES:
Lenth of stay ICU | 15 days
  Time for discharge from the ICU
Days of Mechanical Ventilation | 15 days
  Number of days with ventilatory support
Suplemental Oxigen support | 15 days
  Number of days with need of oxigen suport without Mechanical Ventilation
Viral Load by RT-PCR | 15 days
  changes in viral load
Inflamatory biomarkers | 15 days
  changes in pro- inflamatory and anti-inflamatory biomarkes (IL-6, PCR, Ferritine, D Dimer, IL-8 IL-10
SOFA (sequencial Organ Failure Assesment) | 15 days
  changes in SOFA scale

CONTACTS AND LOCATIONS:
Overall Officials: ORLANDO CARILLO-TORRES, PHD, Study Chair — Hospital General de Mexico Dr. Eduardo Liceaga
Locations (2):
- Mexico (2):
  - Hospital Nava de Alta Especialidad, Mexico City
  - Hospital General de Mexico Dr Eduardo Liceaga, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared by petition.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months after completion up to five years
Access Criteria: proposal should be directed to gmemiinv@gmails.com, to gain access, requestor will need to sign a data access agreement

REFERENCES:
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] Lu H. Drug treatment options for the 2019-new coronavirus (2019-nCoV). Biosci Trends. 2020 Mar 16;14(1):69-71. doi: 10.5582/bst.2020.01020. Epub 2020 Jan 28. PMID 31996494
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] van Griensven J, Edwards T, de Lamballerie X, Semple MG, Gallian P, Baize S, Horby PW, Raoul H, Magassouba N, Antierens A, Lomas C, Faye O, Sall AA, Fransen K, Buyze J, Ravinetto R, Tiberghien P, Claeys Y, De Crop M, Lynen L, Bah EI, Smith PG, Delamou A, De Weggheleire A, Haba N; Ebola-Tx Consortium. Evaluation of Convalescent Plasma for Ebola Virus Disease in Guinea. N Engl J Med. 2016 Jan 7;374(1):33-42. doi: 10.1056/NEJMoa1511812. PMID 26735992
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066